CLINICAL TRIAL: NCT00349141
Title: A Phase I/II Dose Escalation Study of a Vero Cell-Derived, Whole Virus H5N1 Influenza Vaccine in Healthy Volunteers Aged 18 to 45 Years
Brief Title: Safety and Immunogenicity Study of an Inactivated H5N1 Influenza Vaccine (Whole Virion, Vero Cell Derived)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 810501
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2007-10

CONDITIONS: Influenza
Keywords: Pandemic influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Whole virion, Vero cell-derived influenza vaccine containing H5N1 HA antigen

SUMMARY:
The objective of this study is to assess the safety and immunogenicity of 4 different doses of adjuvanted and non-adjuvanted mock-up pandemic influenza vaccine. Subjects will be enrolled sequentially into 3 study cohorts with 4 escalating doses of H5N1 hemagglutininin antigen (3.75 µg adjuvanted, 7.5 µg adjuvanted/non-adjuvanted, 15 µg adjuvanted/non-adjuvanted, 30 µg adjuvanted). Starting with the lowest dose level, subjects will receive 2 vaccinations (21 days apart) at the dose to which they were assigned. Subjects will be monitored for safety and for antibody response to the vaccine. A data safety monitoring board will review and evaluate all the safety data obtained for a dose level before allowing administration of the next (higher) dose.

ELIGIBILITY:
Inclusion Criteria:

Male and femal subjects who

* are 18 to 45 years of age, inclusive, on the day of screening;
* have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry;
* are clinically healthy, as determined by medical history and physical examination;
* agree to keep a daily record of symptoms;
* if female and capable of bearing children, have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Subjects who

* are at high risk of contracting H5N1 influenza infection (e.g. poultry workers);
* suffer from a significant neurological, cardiac, pulmonary (including asthma), hepatic, rheumatic, autoimmune, hematological or renal disorder;
* are unable to lead an independent life as a result of either physical or mental handicap;
* suffer from any kind of immunodeficiency;
* suffer from a disease or are undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs;
* have a history of inflammatory or degenerative neurological disease (e.g. Guillain Barré);
* have a history of severe allergic reactions or anaphylaxis;
* have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating;
* have received a blood transfusion or immunoglobulins within 90 days of study entry;
* have donated blood or plasma within 30 days of study entry;
* have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study;
* have undergone systemic corticoid therapy within 30 days prior to study entry;
* have a functional or surgical asplenia;
* have a known or suspected problem with alcohol or drug abuse;
* were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product;
* are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator;
* if female, are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Principal Investigator — Baxter Healthcare Corporation
Locations (3):
- University Hospital, Department of Clinical Pharmacology, General Hospital Vienna, Vienna, Austria
- Singapore (2):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore

REFERENCES:
- [Derived] Ehrlich HJ, Muller M, Oh HM, Tambyah PA, Joukhadar C, Montomoli E, Fisher D, Berezuk G, Fritsch S, Low-Baselli A, Vartian N, Bobrovsky R, Pavlova BG, Pollabauer EM, Kistner O, Barrett PN; Baxter H5N1 Pandemic Influenza Vaccine Clinical Study Team. A clinical trial of a whole-virus H5N1 vaccine derived from cell culture. N Engl J Med. 2008 Jun 12;358(24):2573-84. doi: 10.1056/NEJMoa073121. PMID 18550874